CLINICAL TRIAL: NCT07316686
Title: Phase I Study of Docetaxel and 177-Lutetium-PSMA-I&T in First-Line Treatment for Patients With Metastatic Castration-Resistant Prostate Adenocarcinoma
Acronym: Lutécio
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP2028
Record Dates: First submitted 2025-09-26; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: A classic 3+3 dose-escalation design will be used to sequentially assign participants to escalating dose levels of docetaxel combined with fixed-dose 177Lu-PSMA-I&T.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Docetaxel 50 mg/m² + 177Lu-PSMA-I&T (Experimental): Patients will receive docetaxel 50 mg/m² IV every 3 weeks plus 177Lu-PSMA-I&T 7.4 GBq IV every 6 weeks. all patients will continue androgen deprivation therapy.
  Interventions: Drug: Docetaxel 50mg/m2; Radiation: 177Lu-PSMA-I&T
- Docetaxel 60 mg/m² + 177Lu-PSMA-I&T (Experimental): Patients will receive docetaxel 60 mg/m² IV every 3 weeks plus 177Lu-PSMA-I&T 7.4 GBq IV every 6 weeks. all patients will continue androgen deprivation therapy.
  Interventions: Drug: Docetaxel 60mg/m2; Radiation: 177Lu-PSMA-I&T
- Docetaxel 75 mg/m² + 177Lu-PSMA-I&T (Experimental): Patients will receive docetaxel 75 mg/m² IV every 3 weeks plus 177Lu-PSMA-I&T 7.4 GBq IV every 6 weeks. all patients will continue androgen deprivation therapy.
  Interventions: Drug: Docetaxel 75 mg/m²; Radiation: 177Lu-PSMA-I&T

INTERVENTIONS:
Drug: Docetaxel 50mg/m2 — Intravenous, 50 mg/m², every 3 weeks, up to 10 cycles
  Arms: Docetaxel 50 mg/m² + 177Lu-PSMA-I&T
Drug: Docetaxel 60mg/m2 — Intravenous, 60 mg/m², every 3 weeks, up to 10 cycles
  Arms: Docetaxel 60 mg/m² + 177Lu-PSMA-I&T
Drug: Docetaxel 75 mg/m² — Intravenous, 75 mg/m², every 3 weeks, up to 10 cycles
  Arms: Docetaxel 75 mg/m² + 177Lu-PSMA-I&T
Radiation: 177Lu-PSMA-I&T — Intravenous administration at a fixed dose of 7.4 GBq every 6 weeks, up to 4 cycles.

SUMMARY:
This is a Phase I, open-label, single-center study evaluating the safety, tolerability, and recommended Phase II dose of docetaxel when combined with a fixed dose of 177-Lutetium-PSMA-I&T in chemotherapy-naïve patients with metastatic castration-resistant prostate cancer (mCRPC). Patients will receive standard androgen deprivation therapy, docetaxel at escalating doses (50 mg/m², 60 mg/m², 75 mg/m² every 3 weeks), and 177Lu-PSMA-I&T at a fixed dose of 7.4 GBq every 6 weeks (up to 4 cycles). A 3+3 dose escalation design will be employed. Secondary endpoints include safety profile, treatment-limiting toxicities, treatment completion rate, and delayed toxicity. Exploratory endpoints include PSA response, radiographic progression-free survival (rPFS), and PERCIST-based response rate.

DETAILED DESCRIPTION:
This is a Phase I, open-label, single-center study designed to evaluate the safety, tolerability, and to determine the recommended Phase II dose (RP2D) of docetaxel when combined with a fixed dose of 177Lu-PSMA-I&T in patients with metastatic castration-resistant prostate cancer (mCRPC) who have not previously received chemotherapy for castration-resistant disease.

All participants will continue receiving androgen deprivation therapy (ADT) throughout the study. The treatment regimen includes docetaxel administered intravenously every 3 weeks at escalating doses of 50 mg/m², 60 mg/m², and 75 mg/m² (up to 10 cycles), combined with 177Lu-PSMA-I&T at a fixed dose of 7.4 GBq every 6 weeks, for up to 4 cycles. A traditional 3+3 dose-escalation design will be used, allowing sequential patient enrollment and assessment of dose-limiting toxicities (DLTs) during the first 3 weeks to establish the optimal docetaxel dose for future studies.

Treatment will continue until completion of 10 cycles of docetaxel and 4 cycles of 177Lu-PSMA-I&T, or until disease progression, unacceptable toxicity, or withdrawal of consent. Imaging exams, including SPECT, will be performed after each lutetium administration for dosimetry assessment.

The primary endpoint is the determination of the RP2D of docetaxel when combined with 177Lu-PSMA-I&T. Secondary endpoints include evaluation of the overall safety profile, incidence of DLTs, treatment completion rate, and monitoring of late toxicities. Exploratory endpoints include PSA response (≥50% decline), radiographic progression-free survival (rPFS), and response rate based on PERCIST criteria using PSMA-PET.

Patients will undergo imaging assessments every 6 weeks (±7 days), including PSMA-PET/CT, FDG-PET/CT, CT scans, and bone scintigraphy. Laboratory tests will be performed every 3 weeks during treatment and every 6 weeks during the post-treatment follow-up, for up to 24 weeks.

Key inclusion criteria include: male patients aged 18 years or older, histologically confirmed adenocarcinoma of the prostate, documented metastatic disease by conventional imaging, castration-resistant disease with testosterone levels <50 ng/mL, ECOG performance status of 0-1, adequate organ function, and positive 68Ga-PSMA-PET/CT uptake according to protocol-defined parameters.

Key exclusion criteria include: presence of small-cell or neuroendocrine tumor components, prior chemotherapy or radiopharmaceuticals for castration-resistant disease, recent or active second malignancies, significant discordance between FDG-PET/CT and PSMA-PET/CT, visible brain metastases, severe urinary incontinence, or any clinical condition that, in the investigator's judgment, would contraindicate the use of docetaxel or 177Lu-PSMA-I&T. Full details of inclusion and exclusion criteria are provided in the study protocol.

This study aims to establish the optimal dose of docetaxel in combination with 177Lu-PSMA-I&T and to generate preliminary safety and efficacy data for treating patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 years or older.
2. Histological or cytological diagnosis of prostate adenocarcinoma. The presence of intraductal or cribriform carcinoma will be allowed.
3. Presence of metastatic disease on conventional imaging exams (bone scintigraphy and/or CT scan or MRI).
4. Patients with castration-resistant disease, defined as testosterone <50 ng/mL in the context of prior orchiectomy or ongoing androgen deprivation therapy (ADT) with LHRH agonists or antagonists, plus at least one of the criteria below:
5. PSA ≥2.0 ng/mL with at least two consecutive PSA rises at intervals of at least 1 week.
6. Radiologic progression defined by the investigator.
7. Clinical progression defined by the investigator.
8. Performance status per the Eastern Cooperative Oncology Group (ECOG) equal to 0 or 1.
9. Willingness to continue ongoing ADT.
10. Adequate organ function as defined below:

    * Parameter Requirement
    * Neutrophils ≥ 1,500/µL
    * Hemoglobin ≥ 12 g/dL
    * Platelets ≥ 100,000/µL
    * Creatinine ≤ 1.5 x upper limit of normal
    * Potassium > 3.5 mmol/L and <5.0 mmol/L
    * Total Bilirubin ≤ ULN (unless Gilbert's disease)
    * AST (TGO) ≤ 2.5 x ULN
    * ALT (TGP) ≤ 2.5 x ULN
11. 68Ga-PSMA-PET/CT performed during the screening phase showing metastatic (extraprosthetic and extrapelvic) disease with radiotracer uptake and:
12. SUVmax ≥20 in at least one site;
13. SUVmax >10 in all other measurable metastatic sites.
14. Lesions with uptake at least 1.5 times greater than hepatic background will be considered measurable.

Exclusion Criteria:

1. Presence of any small-cell or neuroendocrine component of prostate carcinoma.
2. Prior receipt of chemotherapy or radiopharmaceuticals in the castration-resistant setting.
3. Presence of another active malignancy requiring treatment or a cancer diagnosis within the past 5 years. Carcinoma in situ of any site, squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or papillary bladder tumors will be allowed if previously treated.
4. Severe urinary incontinence at the investigator's discretion.
5. 18F-FDG-PET/CT will be performed during screening and will be considered exclusionary if there is discordance with the 68Ga-PSMA-PET/CT. Discordance is defined as FDG-hypermetabolic lesions with absent or low PSMA uptake (SUVmax <10) in more than 50% of measurable metastatic lesions.
6. Patients with brain metastases visible on 68Ga-PSMA-PET/CT.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) of docetaxel in combination with 177Lu-PSMA-I&T | First 3 weeks
  Determination of the recommended Phase II dose using a standard 3+3 dose-escalation design.

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | first 3 weeks.
  Incidence of dose-limiting toxicities (DLTs)
Overall safety profile (CTCAE v5.0) | Up to 24 weeks
  Overall safety profile (CTCAE v5.0)
Treatment completion rate | Up to 24 weeks
  Treatment completion rate (≥4 doses of lutetium and ≥7 doses of docetaxel)
Incidence of late toxicities | Up to 24 weeks post-treatment
  Incidence of late toxicities

OTHER OUTCOMES:
PSA50 response rate | Up to 24 weeks
  PSA50 response rate (≥50% decline from baseline)
Radiographic progression-free survival (rPFS) per PCWG3 | Up to 12 months
  Radiographic progression-free survival (rPFS) per PCWG3
PERCIST-based response rate via PSMA-PET | Up to 12 months
  PERCIST-based response rate via PSMA-PET

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Buchpiguel, MD, PhD, Study Director — Full Professor, Department of Radiology and Oncology; José Mauricio Mota, MD, PhD, Principal Investigator — Medical oncology
Locations (1):
- Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It has been decided not to share individual participant data (IPD) related to the study for several reasons. Protecting the privacy of participants is a priority.
  Sharing IPD may expose sensitive information that, even when de-identified, can be traced back to individuals. Furthermore, the complexity of the data makes sharing challenging without the risk of misunderstandings or misinterpretations, which could compromise the integrity of the research. Sharing IPD without the explicit consent of participants may violate ethical principles of respect and protection. There is also a need to comply with regulatory guidelines governing data sharing to avoid potential legal issues. Finally, the focus will be on disseminating aggregated results that can benefit the scientific community and the public without compromising individual privacy.

REFERENCES:
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] INSTITUTO NACIONAL DO CÂNCER. Estatísticas de câncer. Disponível em: <https://www.inca.gov.br/numeros-de-cancer>. Acesso em: 4 mar. 2021.
- [Background] Tagawa ST, Milowsky MI, Morris M, Vallabhajosula S, Christos P, Akhtar NH, Osborne J, Goldsmith SJ, Larson S, Taskar NP, Scher HI, Bander NH, Nanus DM. Phase II study of Lutetium-177-labeled anti-prostate-specific membrane antigen monoclonal antibody J591 for metastatic castration-resistant prostate cancer. Clin Cancer Res. 2013 Sep 15;19(18):5182-91. doi: 10.1158/1078-0432.CCR-13-0231. Epub 2013 May 28. PMID 23714732
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Scher HI, Solo K, Valant J, Todd MB, Mehra M. Prevalence of Prostate Cancer Clinical States and Mortality in the United States: Estimates Using a Dynamic Progression Model. PLoS One. 2015 Oct 13;10(10):e0139440. doi: 10.1371/journal.pone.0139440. eCollection 2015. PMID 26460686
- [Background] Scher HI, Heller G. Clinical states in prostate cancer: toward a dynamic model of disease progression. Urology. 2000 Mar;55(3):323-7. doi: 10.1016/s0090-4295(99)00471-9. No abstract available. PMID 10699601
- [Background] Ryan CJ, Smith MR, Fizazi K, Saad F, Mulders PF, Sternberg CN, Miller K, Logothetis CJ, Shore ND, Small EJ, Carles J, Flaig TW, Taplin ME, Higano CS, de Souza P, de Bono JS, Griffin TW, De Porre P, Yu MK, Park YC, Li J, Kheoh T, Naini V, Molina A, Rathkopf DE; COU-AA-302 Investigators. Abiraterone acetate plus prednisone versus placebo plus prednisone in chemotherapy-naive men with metastatic castration-resistant prostate cancer (COU-AA-302): final overall survival analysis of a randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2015 Feb;16(2):152-60. doi: 10.1016/S1470-2045(14)71205-7. Epub 2015 Jan 16. PMID 25601341
- [Background] Rahbar K, Ahmadzadehfar H, Kratochwil C, Haberkorn U, Schafers M, Essler M, Baum RP, Kulkarni HR, Schmidt M, Drzezga A, Bartenstein P, Pfestroff A, Luster M, Lutzen U, Marx M, Prasad V, Brenner W, Heinzel A, Mottaghy FM, Ruf J, Meyer PT, Heuschkel M, Eveslage M, Bogemann M, Fendler WP, Krause BJ. German Multicenter Study Investigating 177Lu-PSMA-617 Radioligand Therapy in Advanced Prostate Cancer Patients. J Nucl Med. 2017 Jan;58(1):85-90. doi: 10.2967/jnumed.116.183194. Epub 2016 Oct 20. PMID 27765862
- [Background] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Background] Nilsson S, Larsen RH, Fossa SD, Balteskard L, Borch KW, Westlin JE, Salberg G, Bruland OS. First clinical experience with alpha-emitting radium-223 in the treatment of skeletal metastases. Clin Cancer Res. 2005 Jun 15;11(12):4451-9. doi: 10.1158/1078-0432.CCR-04-2244. PMID 15958630
- [Background] Hofman MS, Emmett L, Sandhu S, Iravani A, Joshua AM, Goh JC, Pattison DA, Tan TH, Kirkwood ID, Ng S, Francis RJ, Gedye C, Rutherford NK, Weickhardt A, Scott AM, Lee ST, Kwan EM, Azad AA, Ramdave S, Redfern AD, Macdonald W, Guminski A, Hsiao E, Chua W, Lin P, Zhang AY, McJannett MM, Stockler MR, Violet JA, Williams SG, Martin AJ, Davis ID; TheraP Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group. [177Lu]Lu-PSMA-617 versus cabazitaxel in patients with metastatic castration-resistant prostate cancer (TheraP): a randomised, open-label, phase 2 trial. Lancet. 2021 Feb 27;397(10276):797-804. doi: 10.1016/S0140-6736(21)00237-3. Epub 2021 Feb 11. PMID 33581798
- [Background] Heck MM, Tauber R, Schwaiger S, Retz M, D'Alessandria C, Maurer T, Gafita A, Wester HJ, Gschwend JE, Weber WA, Schwaiger M, Knorr K, Eiber M. Treatment Outcome, Toxicity, and Predictive Factors for Radioligand Therapy with 177Lu-PSMA-I&T in Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2019 Jun;75(6):920-926. doi: 10.1016/j.eururo.2018.11.016. Epub 2018 Nov 22. PMID 30473431
- [Background] Fizazi K, Scher HI, Molina A, Logothetis CJ, Chi KN, Jones RJ, Staffurth JN, North S, Vogelzang NJ, Saad F, Mainwaring P, Harland S, Goodman OB Jr, Sternberg CN, Li JH, Kheoh T, Haqq CM, de Bono JS; COU-AA-301 Investigators. Abiraterone acetate for treatment of metastatic castration-resistant prostate cancer: final overall survival analysis of the COU-AA-301 randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2012 Oct;13(10):983-92. doi: 10.1016/S1470-2045(12)70379-0. Epub 2012 Sep 18. PMID 22995653
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Dash A, Pillai MR, Knapp FF Jr. Production of (177)Lu for Targeted Radionuclide Therapy: Available Options. Nucl Med Mol Imaging. 2015 Jun;49(2):85-107. doi: 10.1007/s13139-014-0315-z. Epub 2015 Feb 17. PMID 26085854
- [Background] Beer TM, Armstrong AJ, Rathkopf D, Loriot Y, Sternberg CN, Higano CS, Iversen P, Evans CP, Kim CS, Kimura G, Miller K, Saad F, Bjartell AS, Borre M, Mulders P, Tammela TL, Parli T, Sari S, van Os S, Theeuwes A, Tombal B. Enzalutamide in Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer: Extended Analysis of the Phase 3 PREVAIL Study. Eur Urol. 2017 Feb;71(2):151-154. doi: 10.1016/j.eururo.2016.07.032. Epub 2016 Jul 28. PMID 27477525